CLINICAL TRIAL: NCT03372720
Title: Fractional CO2 Laser Therapy for Survivors of Gynecologic Malignancies
Brief Title: Fractional CO2 Laser Therapy in Minimizing Genitourinary Syndrome of Menopause in Gynecological Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Allison Quick, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-17261; NCI-2017-02051 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-11-13; First posted 2017-12-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Cervical Carcinoma; Dyspareunia; Endometrial Carcinoma; Ovarian Carcinoma; Vaginal Carcinoma; Vaginal Dryness; Vulvar Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Dyspareunia; Endometrial Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (fractional CO2 laser therapy) (Experimental): Patients undergo fractional CO2 laser therapy at 3 time points 30 days apart.
  Interventions: Procedure: Laser Therapy; Other: Questionnaire Administration
- Arm II (sham laser therapy) (Sham Comparator): Patients undergo sham laser therapy at 3 time points 30 days apart. Patients may then crossover to Arm I.
  Interventions: Other: Questionnaire Administration; Procedure: Sham Intervention

INTERVENTIONS:
Procedure: Laser Therapy — Undergo fractional CO2 laser therapy
  Other Names: Therapy, Laser
  Arms: Arm I (fractional CO2 laser therapy)
Other: Questionnaire Administration — Ancillary studies
Procedure: Sham Intervention — Undergo sham laser therapy
  Arms: Arm II (sham laser therapy)

SUMMARY:
This randomized pilot trial studies how well fractional carbon dioxide (CO2) laser therapy works in minimizing genitourinary syndrome of menopause (GSM) in gynecological cancer survivors. Fractional CO2 laser therapy may reduce symptoms of GSM in survivors of gynecologic cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a pilot trial to estimate the proportion of gynecologic cancer patients with vaginal dryness or dyspareunia, who will have an improvement in their symptoms with vaginal laser therapy compared to sham treatment based on the Vaginal Assessment Scale (VAS).

SECONDARY OBJECTIVES:

I. To evaluate toxicity associated with vaginal laser therapy in this population.

II. To determine how many women with the defined patient eligibility will complete all treatments.

III. To determine the feasibility of the crossover design for potential use in a phase III trial.

IV. To determine improvement in objective findings of vaginal atrophy with vaginal laser therapy versus sham treatment.

V. To determine improvement in sexual function as measured by Female Sexual Function Index (FSFI), Female Sexual Distress Scale-Revised (FSDS), and scales for sexual satisfaction and behavior with vaginal laser therapy versus sham treatment.

VI. To determine improvement in urinary symptoms of urogenital atrophy with vaginal laser therapy versus sham treatment using the Urogenital Distress Inventory (UDI).

VII. To demonstrate satisfaction with vaginal fractional CO2 laser therapy.

OUTLINE: Patients are randomized in to 1 of 2 arms.

ARM I: Patients undergo fractional CO2 laser therapy at 3 time points 30 days apart.

ARM II: Patients undergo sham laser therapy at 3 time points 30 days apart. Patients may then crossover to Arm I.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Women with cervical, endometrial, vaginal, vulvar or ovarian cancer who have completed all cancer related treatment >= 6 months prior to enrollment

  * Any form of hysterectomy, including radical hysterectomy permitted
  * Must have no evidence of recurrent disease on pelvic exam within past 3 months
  * Radiation therapy is permitted but not required
* Patient reported dyspareunia and/or vaginal dryness with severity of >= 4 on a scale from 0 (none) to 10 (most severe) that has been persistent over >= 4 weeks and/or the inability to be sexually active due to pain

Exclusion Criteria:

* Patients with recurrent or metastatic endometrial, vaginal, vulvar, cervical, or ovarian cancer
* Pelvic organ prolapse stage II or higher
* Prior reconstructive pelvic surgery involving mesh
* Hormone replacement therapy or vaginal estrogen therapy within 6 weeks prior to enrollment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Change in genitourinary syndrome of menopause (GSM) symptoms | Baseline to 12 weeks
  Will be assessed by the Vaginal Assessment Scale (VAS). Will be summarized and compared between the treatment arms using a two-sample t-test or a Wilcoxon rank sum test, with a two-sided alternative for each. Will also analyze this endpoint graphically by plotting the VAS scores through time by treatment arm. Additionally, will correlate the scores from the VAS with other validated measures using a Spearman's correlation coefficient in an exploratory manner.

SECONDARY OUTCOMES:
Feasibility as measured by number of patients able to complete 3 study visitis | Up to 1 month
  A crossover design to determine the feasibility of the crossover design for potential use in a phase III trial by summarizing the proportion of patients who are unable to tolerate the study treatment prior to completing the 3 treatments
Improvement in objective findings of vaginal atrophy | Up to 1 month
  Will determine improvement in objective findings of vaginal atrophy with vaginal laser therapy versus sham treatment.
Improvement in sexual function by FSFI | Up to 1 year
  Will determine improvement in sexual function as measured by Female Sexual Function Index (FSFI)
Improvement in sexual function FSDS | Up to 1 year
  Will determine improvement in sexual function as measured by Female Sexual Distress Scale-Revised (FSDS)
Improvement in urinary symptoms | Up to 1 month
  Will determine improvement in urinary symptoms of urogenital atrophy with vaginal laser therapy versus sham treatment using the Urogenital Distress Inventory (UDI). The change in dyspareunia and dryness between baseline (T0) and T4 will be calculated and compared between the treatment and sham arms using a two sample t-test or Wilcoxon rank sum test.
Incidence of adverse events | Up to 1 month
  Adverse event grading will be done according to the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE)
Number of patients complete all treatments | Up to 1 month
  Summarize the proportion of patients who are able to tolerate the study treatment and complete the 3 treatments.
Satisfaction with vaginal fractional CO2 laser therapy | Up to 1 month
  Patients will be asked to rate their satisfaction with the procedure on a likert-type scale of 1-10 with 1 being completely dissatisfied and 10 being extremely satisfied. Participants will be asked to rate their satisfaction on this scale after each treatment and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Quick, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601
- [Derived] Quick AM, Dockter T, Le-Rademacher J, Salani R, Hudson C, Hundley A, Terstriep S, Streicher L, Faubion S, Loprinzi CL, Coleman JS, Wang KC, Lustberg M. Pilot study of fractional CO2 laser therapy for genitourinary syndrome of menopause in gynecologic cancer survivors. Maturitas. 2021 Feb;144:37-44. doi: 10.1016/j.maturitas.2020.10.018. Epub 2020 Dec 2. PMID 33358206
- See also: The Jamesline — http://cancer.osu.edu